CLINICAL TRIAL: NCT02179749
Title: Glucocorticoid Antagonist Treatment of Alcohol Use Disorder
Brief Title: Mifepristone Treatment of Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Scripps Research Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01AA023152 (NIH)
Record Dates: First submitted 2014-06-26; First posted 2014-07-02 (Estimated); Results first posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Alcohol Dependence; Alcohol Use Disorders; Alcohol Abuse; Alcoholism
Keywords: Alcohol-Related Disorders; Substance-Related Disorders; Mental Disorders; Mifepristone; Glucocorticoid Antagonists; Alcohol Treatment; Alcohol
MeSH Terms: conditions — Alcoholism; Alcohol-Related Disorders; Substance-Related Disorders; Mental Disorders | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: mifepristone 1200 mg daily (Active Comparator): 1200 mg mifepristone daily for 1-week given in conjunction with 8 weeks of standardized behavioral therapy
  Interventions: Drug: Mifepristone 1200 mg daily; Behavioral: Standardized behavioral therapy
- Placebo daily, 1-week (Placebo Comparator): Placebo pills daily for 1-week given in conjunction with 8 weeks of standardized behavioral therapy
  Interventions: Behavioral: Standardized behavioral therapy; Drug: Placebo

INTERVENTIONS:
Drug: Mifepristone 1200 mg daily — Mifepristone, 300 mg tablets, Four tablets daily/am for 1-week duration.
  Other Names: Korlym
  Arms: Experimental: mifepristone 1200 mg daily
Behavioral: Standardized behavioral therapy — Standardized behavioral therapy 1 time per week for 8 week duration.
  Other Names: Manually-guided therapy
Drug: Placebo — Placebo tablets, Four tablets daily/am for 1-week duration.
  Other Names: Placebo Comparator
  Arms: Placebo daily, 1-week

SUMMARY:
This is an 8-week, randomized, double-blind, placebo-controlled, 2 arm, parallel groups, study of 1-week of treatment with mifepristone (0, 1200 mg/d) given in conjunction with 8 weeks of manual-guided counseling, and a follow-up visit at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers, 18-65 years of age
* Meets Diagnostic and Statistical Manual (DSM)-V criteria for current alcohol use disorder of moderate or greater severity, defined by DSM-V as ≥ 4 symptoms
* Abstinent a minimum of 3 days (but not more than 30 days) prior to randomization
* In acceptable health in the judgment of the study physician, on the basis of interview, medical history, physical exam, ECG, urine test and lab tests
* Females with childbearing potential must have a negative serum pregnancy test on the screening visit and a negative urine pregnancy test at randomization and agree to use non-hormonal effective birth control for the study duration and one month thereafter

Exclusion Criteria:

* A medical condition or chronic use of a medication that contraindicates the administration of mifepristone
* Significant medical disorders or clinically significant findings on ECG (e.g., prolongation of the corrected QT interval,urine or blood tests that increase potential risk or interfere with study participation as determined by the Study Physician. Note: serum potassium below the normal range must be replaced to normal prior to randomization; individuals with serum potassium outside the range of normal will not be randomized
* Liver function tests more than 3 times the upper limit of normal or elevated bilirubin
* Female subjects with childbearing potential who are pregnant, nursing, or refuse to use effective non hormonal birth control for the 1-week of medication administration and one month thereafter
* Meets Diagnostic and Statistical Manual -V criteria for a major Axis I disorder including mood or anxiety disorders or substance use disorders other than alcohol or nicotine use disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-09; Primary Completion 2019-11 (Actual); Study Completion 2019-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Mason, Ph.D, Principal Investigator — The Scripps Research Institute
Locations (1):
- The Scripps Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited for study participation at the Laboratory of Clinical Psychopharmacology at The Scripps Research Institute in La Jolla, CA from 10/13/2014-11/6/2019. One Hundred three subjects were enrolled, One Hundred one subjects completed 1-week of medication/placebo, Ninety subjects completed 8-weeks of counseling, and Eighty-four subjects completed a 12-week follow up visit.
Pre-assignment Details: Seventy-one subjects were excluded prior to enrollment: sixty-seven did not meet admission criteria and four declined to participate.
Groups:
- Experimental: Mifepristone 600 mg Day: 600 mg mifepristone daily for 1-week given in conjunction with 8 weeks of standardized behavioral therapy
  Mifepristone 600 mg daily: Mifepristone, 300 mg tablets, Four tablets daily/am (Two 300 mg and two placebo tablets) for 1-week duration.
  Standardized behavioral therapy: Standardized behavioral therapy 1 time per week for 8 week duration.
Period: Overall Study
Arm/Group | Experimental: Mifepristone 1200 mg Daily | Placebo Daily, 1-week | Experimental: Mifepristone 600 mg Day
Started | 49 | 32 | 22
Completed | 49 | 32 | 20
Not Completed | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Daily, 1-week: Placebo pills daily for 1-week given in conjunction with 8 weeks of standardized behavioral therapy
  . Placebo: Placebo tablets, Four tablets daily/am for 1-week duration.
  Standardized behavioral therapy: Standardized behavioral therapy 1 time per week for 8 week duration
- Total: Total of all reporting groups
Arm/Group | Experimental: Mifepristone 1200 mg Daily | Placebo Daily, 1-week | Experimental: Mifepristone 600 mg Day | Total
Number analyzed (Participants) | 49 | 32 | 22 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (11.0) | 46.4 (11.9) | 44.4 (12.3) | 46.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 8 | 38
  Male | 32 | 19 | 14 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 4 | 22
  Not Hispanic or Latino | 39 | 24 | 18 | 81
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 3
  White | 38 | 27 | 17 | 82
  More than one race | 4 | 4 | 2 | 10
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 49 | 32 | 22 | 103
DSM-V symptom count [Mean (Standard Deviation); unit: symptoms] | 8.63 (1.53) | 8.22 (1.99) | 8.59 (2.30) | 8.5 (1.86)

OUTCOME MEASURES:

1. Primary Outcome: Drinking Quantity Per Day
Description: Drinking quantity in standard drinks per day is measured by the Timeline Followback interview.
  A standard drink contains 14 grams of alcohol, e.g., 1.5 ounces of distilled spirits, 5 ounces of wine, or 12 ounces of beer.
Time Frame: Participants will be followed for up to 12 weeks post-assignment
Population: Individuals with moderate or greater severity level of alcohol use disorder.
Measure: Mean (Standard Error); unit: Standard drinks per day
Groups:
- Placebo; 600 mg/d of Mifepristone; 1200 mg/d of Mifepristone: 1 week of double-blind study medication 8 weeks of counseling
Arm/Group | Placebo | 600 mg/d of Mifepristone | 1200 mg/d of Mifepristone
Number analyzed (Participants) | 32 | 22 | 49
Standard drinks per day | 1.25 (0.21) | 1.38 (0.21) | 1.10 (0.21)
Statistical Analysis 1: Comparison: Placebo vs 600 mg/d of Mifepristone vs 1200 mg/d of Mifepristone; Test type: Superiority; p = 0.51, ANOVA; Mean Difference (Final Values) = 0.52, Standard Error of Mean 0.20
Statistical Analysis 2: Comparison: Placebo vs 600 mg/d of Mifepristone vs 1200 mg/d of Mifepristone; Latent growth model includes one week on study drug and two weeks after the last dose of study drug. Principal predictors were drug plasma concentration and baseline treatment goal of abstinence or non abstinence. Arms were combined for this analysis; Test type: Superiority; p = 0.038, Mixed Models Analysis; Slope = 0.08, Standard Error of Mean .04

2. Secondary Outcome: Craving
Description: Alcohol Craving Questionnaire; minimum value equals 12, maximum value equals 84; higher scores mean greater craving for alcohol.
Time Frame: Participants will be followed for up to 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Experimental: Mifepristone 1200 mg Daily | Placebo Daily, 1-week | Experimental: Mifepristone 600 mg Day
Number analyzed (Participants) | 49 | 32 | 22
score on a scale | 29.02 (36.69) | 33.66 (36.69) | 28.33 (36.69)
Statistical Analysis 1: Comparison: Experimental: Mifepristone 1200 mg Daily vs Placebo Daily, 1-week vs Experimental: Mifepristone 600 mg Day; Test type: Superiority; p = 0.50, ANOVA; 411 and 102 degrees of freedom; Mean Difference (Final Values) = 0.15, Standard Error of Mean 36.7

ADVERSE EVENTS:
Time Frame: Study medication was administered for one week. Adverse event data were collected during this 1-week of medication or placebo treatment. These treatment emergent adverse events were followed until resolution over the 8-week behavioral therapy period.
Arm/Group | Experimental: Mifepristone 1200 mg Daily | Placebo Daily, 1-week | Experimental: Mifepristone 600 mg Day
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/32 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/49 | 1/32 | 0/22
Other Adverse Events (participants affected / at risk) | 17/49 | 8/32 | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Mifepristone 1200 mg Daily (N=49) | Placebo Daily, 1-week (N=32) | Experimental: Mifepristone 600 mg Day (N=22)
Syncope (Nervous system disorders) | 0 | 1 | 0 — Syncope episode while riding a horse resulting in a fall. Overnight hospitalization required.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Mifepristone 1200 mg Daily (N=49) | Placebo Daily, 1-week (N=32) | Experimental: Mifepristone 600 mg Day (N=22)
Headache (Nervous system disorders) | 12 | 4 | 2
Fatigue (Psychiatric disorders) | 5 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Study Protocol -IND (2014-07-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT02179749/Prot_SAP_ICF_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2014-02-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT02179749/SAP_001.pdf
  • Informed Consent Form: Informed Consent (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT02179749/ICF_002.pdf